CLINICAL TRIAL: NCT01099150
Title: Acute Effects of the Consumption of Dark Chocolate Enriched in Flavan-3-ols on Platelet Function and the Platelet Proteome
Brief Title: Dark Chocolate and Platelet Function in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Rural and Environment Research and Analysis Directorate (RERAD, UK) (Unknown); Biotechnology and Biological Sciences Research Council (Other); Natraceutical Industrial S.L.U., Valencia, Spain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 600; 09/002 (Other: Rowett Human Studies Ethical Review Panel)
Record Dates: First submitted 2010-03-25; First posted 2010-04-06 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Disease
Keywords: Platelets; Platelet aggregation; Platelet activation; Platelet function; Light transmission aggregometry; Platelet Function Analyzer-100 (PFA-100); P-selectin; Fibrinogen receptor; Glycoprotein IIb-IIIa; Chocolate; Cocoa; Flavan-3-ols; Procyanidins
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Proanthocyanidins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 42 healthy volunteers - crossover (Experimental): Acute consumption of three interventions (60 g dark chocolate enriched in flavan-3-ols, 60 g standard dark chocolate, or 60 g white chocolate) on three separate days (at least 2 weeks apart) in random order.
  Post-prandial measurements at t = 0 h, t = 2 h and t = 6 h.
  Interventions: Dietary Supplement: Dark chocolate enriched in flavan-3-ols and procyanidins; Dietary Supplement: Standard dark chocolate; Dietary Supplement: White chocolate

INTERVENTIONS:
Dietary Supplement: Dark chocolate enriched in flavan-3-ols and procyanidins — Acute consumption (within 15 minutes) of 60 g of chocolate containing ~900 mg of total flavan-3-ols and procyanidins.
  Other Names: CocoanOX12%-containing chocolate
Dietary Supplement: Standard dark chocolate — Acute consumption (within 15 minutes) of 60 g of chocolate containing ~400 mg total flavan-3-ols and procyanidins.
Dietary Supplement: White chocolate — Acute consumption (within 15 minutes) of 60 g of white chocolate containing no flavan-3-ols and procyanidins.

SUMMARY:
Cardiovascular disease is a major cause of mortality worldwide and responsible for one out of three global deaths. A main characteristic of cardiovascular disease is impaired blood flow and formation of blood clots. Platelets are clot-forming cells responsible for the prevention of bleeding. However, in disease conditions they may be overly activated, promoting blood clots and blockage of blood vessels.

Consumption of diets rich in fruits and vegetables decreases mortality from cardiovascular disease through a number of mechanisms, including the prevention of platelet clotting and aggregation. There is some evidence suggesting that platelet aggregation may be modulated through a group of compounds known as flavan-3-ols, which are found in various foods, and especially in cocoa. However, the mechanisms by which those compounds affect platelet function are not yet fully understood. We designed a human study assessing the mechanisms by which flavan-3-ols from cocoa beneficially affect platelet function and the platelet proteome.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a primary cause of premature deaths worldwide, with incidence rates in the United Kingdom, particularly in Scotland, being amongst the highest worldwide. Thus identification of dietary components that most effectively prevent CVD is potentially of wide public health benefit.

Consumption of diets rich in plant-based products protects against the development of CVD. Such effects have been ascribed in part to polyphenols, which are non-nutritive but, potentially bioactive secondary metabolites ubiquitous found in fruits, vegetables, herbs, spices, teas and wines. The beneficial effects of polyphenols on CVD is believed to be mediated, at least in part, though improving platelet function. At least 10 human intervention studies found a consistent and robust beneficial effect of cocoa products on platelet function, but unfortunately all of these studies used only one or two methods to assess platelet function, therefore only getting limited insights into the complex physiological behavior of platelets. In addition, none of these studies assessed potential mechanisms by which flavan-3-ols may inhibit platelet function. Schramm et al. have shown that consumption of chocolate rich in flavan-3-ols and their oligomers (procyanidins) lead to increased production of prostacyclin, a strong platelet inhibitor. This finding has also been observed when aortic endothelial cells are treated with procyanidins in vitro. Thus the stimulation of prostacyclin production in endothelial cells may reflect one pathway by which flavan-3-ols indirectly inhibit platelet activation. Many other potential mechanisms are discussed in the literature but so far the evidence for such mechanisms is limited or non-existing.

In this study we assess effects of consumption of chocolate enriched in flavan-3-ols on platelet function by measuring not only platelet aggregation, but also in vitro coagulation and platelet activation in healthy humans. In addition, we examine the effects of consumption of flavan-3-ols on the regulation of the platelet proteome to elucidate pathways by which these bioactive cocoa compounds affect platelet function.

HYPOTHESIS

Acute consumption of a moderate amount of dark chocolate enriched in flavan-3-ols results in decreased platelet activation and aggregation by decreasing the levels of thromboxane A2 produced by endothelial cells.

OBJECTIVES

The main objective of the proposed study is to determine whether consumption of 60 g dark chocolate enriched in flavan-3-ols results in decreased platelet activation and aggregation by decreasing levels of thromboxane A2, as well as assessing what other mechanisms could be involved.

The specific objectives of the proposed study are to determine:

1. whether acute intake of 60 g dark chocolate enriched in flavan-3-ols, as compared with standard dark chocolate low in flavan-3-ols and white chocolate containing no flavan-3-ols, affects platelet aggregation, thromboxane A2 formation upon aggregation, in vitro bleeding time, P-selectin expression, and activation of the fibrinogen receptor;
2. whether and how acute intake of 60 g dark chocolate enriched in flavan-3-ols, as compared with standard dark chocolate and white chocolate, affects the platelet proteome, and thereby potential new biomarkers of platelet function, as well as protein levels of anti-oxidant enzymes;
3. identities and concentrations of flavan-3-ols and their metabolites in plasma and/ or urine 2 and 6 h after acute intake of 60 g dark chocolate enriched in flavan-3-ols, as compared with standard dark chocolate and white chocolate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female volunteers, aged between 18 and 70 years

Exclusion Criteria:

Subjects are excluded if:

* they are taking aspirin or aspirin-containing drugs, other anti-inflammatory drugs, or any drugs or herbal medicines known to alter platelet function or the haemostatic system in general (without a minimum washout period of one month)
* they are taking fish oils or evening primrose oil, or fat soluble vitamin supplements within the last 4 weeks
* they are taking any medicine known to affect lipid and/or glucose metabolism
* they are taking hormone replacement therapy
* they have any known clinical signs of diabetes, hypertension, renal, hepatic, hematological disease, gastrointestinal disorders, endocrine disorders, coronary heart disease, infection or cancer
* they are suffering from alcohol or any other substance abuse or are having eating disorders
* they are usually consuming a vegetarian diet
* they have a BMI below 18 or above 35 kg/ sqm
* they are undertaking more than 6 hours of vigorous exercise per week
* they are having an abnormal menstrual cycle
* they are pregnant
* they suffer from an allergy to cocoa or any of the ingredients contained within either of the chocolate bars
* they have been giving a pint of blood for transfusion purposes within the last month
* they have a low platelet count (< 170 x 10E09/ L)
* they have unsuitable veins for blood sampling and/ or cannulation
* their hematocrit is below 40 % for males and 35 % for females
* their haemoglobin is below 130 g/ L for males and 115 g/ L for females
* they are not able to travel on their own to the Rowett Institute of Nutrition and Health, Aberdeen for each of the interventions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in light transmission aggregometry of platelet-rich plasma | Post-prandial, up to 6 hours after chocolate consumption
  * Using a Helena Platelet Aggregation Chromogenic Kinetics System-4 (PACKS-4) light transmission aggregometer
  * Induced by adenosine diphosphate (ADP) and thrombin receptor-activating peptide (TRAP)

SECONDARY OUTCOMES:
Change in ex vivo bleeding time using the Platelet Function Analyzer-100 (PFA-100) | Post-prandial, up to 6 hours after chocolate consumption
  Using collagen-epinephrine coated cartridges.
Change in P-selectin expression and activation of the fibrinogen receptor by flow cytometry | Post-prandial, up to 6 hours after chocolate consumption
  * P-selectin expression as early marker for platelet activation
  * Activated fibrinogen receptor as late marker for platelet activation
  * Induced by ADP and TRAP
  * Using BD FACSArray Bioanalyzer
Levels of flavan-3-ols and their metabolites in plasma and urine | Post-prandial, up to 6 hours after chocolate consumption
  * Using liquid chromatography-tandem mass spectrometry (LC-MS/MS)
  * Enzyme-hydrolysed for total flavan-3-ols ((-)-epicatechin equivalents)
  * Non-Hydrolysed for metabolic profile
Changes in the platelet proteome | Post-prandial, 2 hours after chocolate ingestion
  Using 2D-gel electrophoresis and LC-MS/MS identification of proteins.
Changes in thromboxane A2 production induced by ADP and TRAP | Post-prandial, up to 6 hours after chocolate consumption
  Using enzyme-linked immunosorbent assay (ELISA) in plasma after platelet aggregation
Levels of prostacyclin and/ or leukotrienes in plasma | Post-prandial, up to 6 hours after chocolate consumption
  Using high performance liquid chromatography (HPLC) and/ or immunoassays
Total phenolics in urine | Post-prandial, up to 6 hours after chocolate consumption
  Using the Folin-Ciocalteu assay
Total catechins in urine | Post-prandial, up to 6 hours after chocolate consumption
  Using an adaption of the DMACA assay
Urinary creatinine | Post-prandial, up to 6 hours after chocolate consumption
  Using a Thermo KONELAB 30 selective chemistry analyser (Thermo Scientific, Hertfordshire, UK) and its respective kit
  To be used for normalisation of urinary flavan-3-ols and total phenolics from spot urine samples.
Analysis of flavan-3-ol and procyanidin contents in study chocolates | At the beginning (April 2009) and end (October 2009) of the intervention period
  Using an HPLC method
Non-targeted 1H-NMR of plasma and urine samples | Post-prandial, up to 6 hours after chocolate consumption
  To establish a metabolic profile - markers of intake and potential effects on host metabolism
Non-targeted LC-MS of urine samples | Post-prandial, just before and 6 hours after chocolate consumption
  To establish a metabolic profile - markers of intake and potential effects on host metabolism
Markers of oxidative stress in plasma | Post-prandial, up to 6 hours after chocolate consumption
  1. Plasma levels of lipid peroxides (thiobarbituric acid-reactive substances, TBARS)
  2. Activity of glutathione peroxidase (Only at t = 2 h after chocolate ingestion)
Fatty acid analysis of study chocolates | Shortly after the intervention period was finished (February 2009)
  Using the fatty acid methyl ester (FAME) analysis and a gas chromatographic approach

CONTACTS AND LOCATIONS:
Overall Officials: Baukje de Roos, MSc PhD, Principal Investigator — University of Aberdeen Rowett Institute of Nutrition and Health
Locations (1):
- University of Aberdeen Rowett Institute of Nutrition and Health, Aberdeen, Aberdeenshire, United Kingdom

REFERENCES:
- [Background] Baba S, Osakabe N, Yasuda A, Natsume M, Takizawa T, Nakamura T, Terao J. Bioavailability of (-)-epicatechin upon intake of chocolate and cocoa in human volunteers. Free Radic Res. 2000 Nov;33(5):635-41. doi: 10.1080/10715760000301151. PMID 11200094
- [Background] Bordeaux B, Yanek LR, Moy TF, White LW, Becker LC, Faraday N, Becker DM. Casual chocolate consumption and inhibition of platelet function. Prev Cardiol. 2007 Fall;10(4):175-80. doi: 10.1111/j.1520-037x.2007.06693.x. PMID 17917513
- [Background] de Roos B, Duthie SJ, Polley AC, Mulholland F, Bouwman FG, Heim C, Rucklidge GJ, Johnson IT, Mariman EC, Daniel H, Elliott RM. Proteomic methodological recommendations for studies involving human plasma, platelets, and peripheral blood mononuclear cells. J Proteome Res. 2008 Jun;7(6):2280-90. doi: 10.1021/pr700714x. Epub 2008 May 20. PMID 18489134
- [Background] Flammer AJ, Hermann F, Sudano I, Spieker L, Hermann M, Cooper KA, Serafini M, Luscher TF, Ruschitzka F, Noll G, Corti R. Dark chocolate improves coronary vasomotion and reduces platelet reactivity. Circulation. 2007 Nov 20;116(21):2376-82. doi: 10.1161/CIRCULATIONAHA.107.713867. Epub 2007 Nov 5. PMID 17984375
- [Background] Guerrero JA, Navarro-Nunez L, Lozano ML, Martinez C, Vicente V, Gibbins JM, Rivera J. Flavonoids inhibit the platelet TxA(2) signalling pathway and antagonize TxA(2) receptors (TP) in platelets and smooth muscle cells. Br J Clin Pharmacol. 2007 Aug;64(2):133-44. doi: 10.1111/j.1365-2125.2007.02881.x. Epub 2007 Apr 10. PMID 17425630
- [Background] Hamed MS, Gambert S, Bliden KP, Bailon O, Singla A, Antonino MJ, Hamed F, Tantry US, Gurbel PA. Dark chocolate effect on platelet activity, C-reactive protein and lipid profile: a pilot study. South Med J. 2008 Dec;101(12):1203-8. doi: 10.1097/SMJ.0b013e31818859eb. PMID 19005437
- [Background] Heptinstall S, May J, Fox S, Kwik-Uribe C, Zhao L. Cocoa flavanols and platelet and leukocyte function: recent in vitro and ex vivo studies in healthy adults. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S197-205; discussion S206-9. doi: 10.1097/00005344-200606001-00015. PMID 16794458
- [Background] Hermann F, Spieker LE, Ruschitzka F, Sudano I, Hermann M, Binggeli C, Luscher TF, Riesen W, Noll G, Corti R. Dark chocolate improves endothelial and platelet function. Heart. 2006 Jan;92(1):119-20. doi: 10.1136/hrt.2005.063362. No abstract available. PMID 16365364
- [Background] Hubbard GP, Wolffram S, de Vos R, Bovy A, Gibbins JM, Lovegrove JA. Ingestion of onion soup high in quercetin inhibits platelet aggregation and essential components of the collagen-stimulated platelet activation pathway in man: a pilot study. Br J Nutr. 2006 Sep;96(3):482-8. PMID 16925853
- [Background] Hubbard GP, Wolffram S, Lovegrove JA, Gibbins JM. Ingestion of quercetin inhibits platelet aggregation and essential components of the collagen-stimulated platelet activation pathway in humans. J Thromb Haemost. 2004 Dec;2(12):2138-45. doi: 10.1111/j.1538-7836.2004.01067.x. PMID 15613018
- [Background] Innes AJ, Kennedy G, McLaren M, Bancroft AJ, Belch JJ. Dark chocolate inhibits platelet aggregation in healthy volunteers. Platelets. 2003 Aug;14(5):325-7. doi: 10.1080/0953710031000123681. PMID 12944249
- [Background] Mavrommatis Y, O'Kennedy N, de Roos B et al. Effect of eicosapentaenoic acid or docosahexaenoic acid intervention on platelet aggregation: does soluble epoxide hydrolase play a role? unpublished, 2010
- [Background] Murphy KJ, Chronopoulos AK, Singh I, Francis MA, Moriarty H, Pike MJ, Turner AH, Mann NJ, Sinclair AJ. Dietary flavanols and procyanidin oligomers from cocoa (Theobroma cacao) inhibit platelet function. Am J Clin Nutr. 2003 Jun;77(6):1466-73. doi: 10.1093/ajcn/77.6.1466. PMID 12791625
- [Background] Nardini M, Natella F, Scaccini C. Role of dietary polyphenols in platelet aggregation. A review of the supplementation studies. Platelets. 2007 May;18(3):224-43. doi: 10.1080/09537100601078083. PMID 17497435
- [Background] Natella F, Nardini M, Belelli F, Pignatelli P, Di Santo S, Ghiselli A, Violi F, Scaccini C. Effect of coffee drinking on platelets: inhibition of aggregation and phenols incorporation. Br J Nutr. 2008 Dec;100(6):1276-82. doi: 10.1017/S0007114508981459. Epub 2008 Apr 28. PMID 18439332
- [Background] Natella F, Nardini M, Virgili F, Scaccini C. Role of dietary polyphenols in the platelet aggregation network - A review of the in vitro studies. Curr Top Nutraceut Res 4(1): 1-22, 2006.
- [Background] Ostertag LM, O'Kennedy N, Kroon PA, Duthie GG, de Roos B. Impact of dietary polyphenols on human platelet function--a critical review of controlled dietary intervention studies. Mol Nutr Food Res. 2010 Jan;54(1):60-81. doi: 10.1002/mnfr.200900172. PMID 20058256
- [Background] Pearson DA, Paglieroni TG, Rein D, Wun T, Schramm DD, Wang JF, Holt RR, Gosselin R, Schmitz HH, Keen CL. The effects of flavanol-rich cocoa and aspirin on ex vivo platelet function. Thromb Res. 2002 May 15;106(4-5):191-7. doi: 10.1016/s0049-3848(02)00128-7. PMID 12297125
- [Background] Rechner AR, Kroner C. Anthocyanins and colonic metabolites of dietary polyphenols inhibit platelet function. Thromb Res. 2005;116(4):327-34. doi: 10.1016/j.thromres.2005.01.002. Epub 2005 Feb 8. PMID 16038718
- [Background] Rein D, Paglieroni TG, Wun T, Pearson DA, Schmitz HH, Gosselin R, Keen CL. Cocoa inhibits platelet activation and function. Am J Clin Nutr. 2000 Jul;72(1):30-5. doi: 10.1093/ajcn/72.1.30. PMID 10871557
- [Background] Schewe T, Sadik C, Klotz LO, Yoshimoto T, Kuhn H, Sies H. Polyphenols of cocoa: inhibition of mammalian 15-lipoxygenase. Biol Chem. 2001 Dec;382(12):1687-96. doi: 10.1515/BC.2001.204. PMID 11843182
- [Background] Schramm DD, Wang JF, Holt RR, Ensunsa JL, Gonsalves JL, Lazarus SA, Schmitz HH, German JB, Keen CL. Chocolate procyanidins decrease the leukotriene-prostacyclin ratio in humans and human aortic endothelial cells. Am J Clin Nutr. 2001 Jan;73(1):36-40. doi: 10.1093/ajcn/73.1.36. PMID 11124747
- [Background] Wang-Polagruto JF, Villablanca AC, Polagruto JA, Lee L, Holt RR, Schrader HR, Ensunsa JL, Steinberg FM, Schmitz HH, Keen CL. Chronic consumption of flavanol-rich cocoa improves endothelial function and decreases vascular cell adhesion molecule in hypercholesterolemic postmenopausal women. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S177-86; discussion S206-9. doi: 10.1097/00005344-200606001-00013. PMID 16794456